CLINICAL TRIAL: NCT05640661
Title: Effects of Terminal Visual Feedback Therapy After Immersive Virtual Reality in Patients With Chronic Shoulder Pain : Mixed-Methods Randomized Clinical Trial
Brief Title: Effects of Terminal Visual Feedback Therapy After Immersive Virtual Reality in Patients With Chronic Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Alejandro Luque-Suarez, Head of Physiotherapy Departament, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMalagaVRi
Record Dates: First submitted 2022-11-16; First posted 2022-12-07 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Shoulder Pain; Movement Disorders
Keywords: Virtual Reality
MeSH Terms: conditions — Shoulder Pain; Movement Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terminal visual feedback therapy plus Immersive Virtual reality (Experimental): Active treatment using Virtual Reality software based on pain education and gamified exercise for gradual exposure to shoulder movement.
  The brief intervention will last 3 sessions of 15 minutes during a week, thus taking a total duration of one week of treatment. Within the intervention will consist of a pill of education in pain neuroscience (PNE) of 1 minute duration, followed by an exposure level that will last 2:30 minutes where a progression will be made in number of ranges of motion and speed. Each session will consist of 2 intervention blocks (PNE + Gradual Exposure pill). The content of the PNE educational pills have been selected according to the objective of the study. Subjects will be recorded through an Ipad Tablet, and after performing the entire intervention a terminal visual feedback therapy will be performed by observation of actions in holocentric vision.
  Interventions: Device: Oculus Quest II
- Immersive Virtual Reality (Active Comparator): Active treatment using Virtual Reality software based on pain education and gamified exercise for gradual exposure to shoulder movement. The game involves visual stimuli and shoulder movement exercises in the shoulder flexion and abduction ranges in real time using immersive glasses located on the head and two controls on both hands. Patients will inhabit an avatar from an egocentric perspective.
  The brief intervention will last 3 sessions of 15 minutes during a week, thus taking a total duration of one week of treatment. Within the intervention will consist of a pill of education in pain neuroscience (PNE) of 1 minute duration, followed by an exposure level that will last 2:30 minutes where a progression will be made in number of ranges of motion and speed. Each session will consist of 2 intervention blocks (PNE + Gradual Exposure pill). The content of the PNE educational pills have been selected according to the objective of the study.
  Interventions: Device: Oculus Quest II

INTERVENTIONS:
Device: Oculus Quest II — active treatment using Virtual Reality software based on pain education and gamified exercise for gradual exposure to shoulder movement. The game involves visual stimuli and shoulder movement exercises in the shoulder flexion and abduction ranges in real time using immersive glasses located on the head and two controls on both hands. Patients will inhabit an avatar from an egocentric perspective.
  During the realization of the exposure with VRi they will be recorded through an Ipad Tablet, and after performing the entire intervention a terminal visual feedback therapy will be performed by observation of actions in holocentric vision.
  Other Names: Immersive Virtual Reality + terminal visual feedback therapy
  Arms: Terminal visual feedback therapy plus Immersive Virtual reality
Device: Oculus Quest II — active treatment using Virtual Reality software based on pain education and gamified exercise for gradual exposure to shoulder movement. The game involves visual stimuli and shoulder movement exercises in the shoulder flexion and abduction ranges in real time using immersive glasses located on the head and two controls on both hands. Patients will inhabit an avatar from an egocentric perspective.
  Other Names: Immersive Virtual Reality
  Arms: Immersive Virtual Reality

SUMMARY:
The goal of this clinical trial is effect of terminal visual feedback therapy following the use of immersive virtual reality(VRi) effects on pain,kinesiophobia, fear of pain, disability, self-efficacy, grip strength and range of motion in motion in people with chronic shoulder pain compare with just VRi. The main question[s] it aims to answer are:

* Can terminal visual feedback therapy following the use of immersive virtual reality software decrease movement-evoked pain in patients with chronic shoulder pain compared with just VRi?
* Can terminal visual feedback therapy following the use of immersive virtual reality software increase shoulder flexion range of motion in patients with chronic shoulder pain compared with just VRi?

Participants will use a visual feedback therapy following the use of immersive virtual reality software compared with just specific VRi software

DETAILED DESCRIPTION:
Studio Design Mixed-methods investigation with Randomized Controlled Clinical Trial (RCT). This protocol follows the indications of the guidelines for Clinical Trial Publications (CONSORT) and will follow the TIDIER check-list for the exhaustive description of the interventions that will be performed.

For the qualitative part, a semi-structured interview will be carried out following the indications proposed in the guide for qualitative research publications (COREQ) Target population Patients with persistent musculoskeletal shoulder pain aged 18-65 years primary chronic musculoskeletal pain, according to the International Classification of Diseases-11 (2019) of the International Association for the Study of Shoulder-related Pain (IASP).

Sample size calculation A total of 11 individuals for each treatment group will allow to detect, in numerical variables, differences between pairs of group means of a corresponding magnitude (Flexion range of motion) at 10 points of the standard deviation, with an effect size of 80% maintaining the type I error at a level of 5%. Taking into account a loss of 10%, it would be necessary to include 12 individuals in each group.

Study variables For the qualitative part of the study, a semi-structured interview will be conducted at the beginning of the study and at the end of it, with the same questions in measurements. The questions have been selected and adapted to the persistent shoulder pain of the clinical interview proposal of O'Sullivan et. Al based on functional cognitive therapy (CFT)

* How safe do you feel doing the things in your life that you value?
* How has pain impacted your life?
* What do you think will happen if you lift your shoulder?
* How do you feel when you lift your shoulder?
* How do you feel about the pain?
* Is pain predictable for you? The interviews will be recorded by the principal investigator in order to analyze patients' beliefs and perceptions regarding their shoulder pain, and if there are changes after the intervention.

Interventions This is a randomized clinical trial (RCT) of 2 parallel groups (ratio 1:1) that will be carried out in the Teaching Assistance Unit (UDA) of the Faculty of Health Science of the University of Malaga (UMA). The study protocol will follow the TIDIER check-list for the exhaustive description of the interventions to be performed and the RCT will conform to the Consolidated Standards of Reporting Testing (CONSORT).

Recruitment: Patients will be recruited by invitation to participate via email to the university community, as well as contact with Family Medicine professionals for the referral of patients who meet the inclusion criteria will be invited to participate in the RCT. Doctors involved in the recruitment process will receive a clinical session to ensure that the selection process is carried out according to the inclusion criteria and that participants do not meet the exclusion criteria.

Patients will receive oral information and a written document (Patient Information Sheet). If the patient is interested in participating in the study, after signing the informed consent, he will be summoned to be evaluated by an external evaluator who will perform the initial assessment. The patient will also receive a revocation sheet in case they decide to leave the study at any time. After the initial assessment, participants will be randomly assigned to one of two study groups (experimental or control).

Randomization After the initial evaluation, each patient will be assigned an alphanumeric code for the identification of each subject, thus respecting their anonymity. To perform the randomization procedure, the principal investigator (PI) will receive a list of the alphanumeric codes of the participants and perform a random assignment using the SPSS statistical package.

Blinding An independent biostatistician will perform the statistical analysis without knowing the treatment performed by each group. The intervention cannot be blinded to the participants or the physiotherapists who perform it, but the physiotherapists who perform the intervention will not participate in the patient assessment process and will not know the previous status of the participants or the objectives of the clinical trial.

Intervention

- Control group: An active treatment using Virtual Reality software based on pain education and gamified exercise for gradual exposure to shoulder movement will be performed. The game involves visual stimuli and shoulder movement exercises in the shoulder flexion and abduction ranges in real time using immersive glasses located on the head and two controls on both hands. Patients will inhabit an avatar from an egocentric perspective.

The brief intervention will last 3 sessions of 15 minutes during a week, thus taking a total duration of one week of treatment. Within the intervention will consist of a pill of education in pain neuroscience (PNE) of 1 minute duration, followed by an exposure level that will last 2:30 minutes where a progression will be made in number of ranges of motion and speed. Each session will consist of 2 intervention blocks (PNE + Gradual Exposure pill). The content of the PNE educational pills have been selected according to the objective of the study.

* Pain as an alarm system
* Protectometer
* Sensory and interpretation component
* The complexity of the body
* Threshold depends on context
* PD, Sensitivity
* Intervention group: the participants randomly assigned to the intervention treatment will perform the same protocol as the control group with the difference that during the realization of the exposure with VRi they will be recorded through an Ipad Tablet, and after performing the entire intervention a terminal visual feedback therapy will be performed by observation of actions in holocentric vision.

Data collection procedure The study protocol will be recorded in Clinicaltrials.gov, prior to data collection.

Who will collect the data: A physiotherapist with experience in managing people with persistent musculoskeletal shoulder pain and training by the research team will be responsible for data collection. The videos obtained for visual feedback therapy will be collected by the physiotherapist performing the intervention.

For semi-structured interviews, they will be recorded by the principal investigator for further analysis and coding.

When data will be collected: Pain variables during movement and range of motion will be measured before the intervention and after the intervention in each treatment session Demographic variables will be collected at the beginning of the study. Finally, the variables of Self-efficacy, Kinesiophobia, Fear of pain and disability will be collected at the beginning of the intervention and at the end of the intervention after the week of treatment.

How the data will be collected: all variables will be measured with the self-reported questionnaires discussed in the table above, since they are validated and reliable measures to assess these factors. The semi-structured views will be collected by an electronic recorder for later analysis by the evaluators.

Data analysis

All data will be evaluated to check the normality of its distribution. The numerical variables will be summarized with means and standard deviations and the categorical ones with percentages. Numerical variables that show a distribution far removed from normal will be transformed to obtain distributions close to normal, or otherwise, they will be summarized by using percentiles. For the graphical representation of the distribution of the numerical variables in each treatment group,box and whisker graphs will be used. To represent categorical variables, pie charts will be used.

In order to test the equality of means for numerical variables, Student's T will be applied if the distributions are not far from normal. Otherwise, the Wilcoxon-Mann-Whitney statistics will be calculated. Depending on the observed response to treatment in numerical variables or the observed change in them, several definitions of success/failure for the treatment outcome in individuals will be built.

Logistic regression models to predict treatment success will be adjusted. These models will include those variables that show a statistically significant relationship with the corresponding outcome variables in the univariate analysis. It shall be considered as statistically significant p-values below 0,05. All models will be adjusted for age, gender, pain intensity and pain duration. These variables will be used as adjustment variables due to their importance as factors associated with chronic pain The analysis of the data will be carried out through the use of statistical software R.

For the qualitative part, it will be analyzed by two physiotherapists experts in persistent musculoskeletal pain based on the analysis of the content (latent) in the interviews of the participants of both groups. For this, a methodology consisting of the following steps will be carried out

1. Transcription of interviews in text
2. Extraction of relevant data to categorize into subtopics and topics.
3. Code the information collected in topics and subtopics.
4. Comparison and relationship of the topics found by both evaluators

Ethical aspects

To be carried out, this study will have to be previously approved by the Research Ethics Committee of the University of Malaga (CEUMA) This study will be guided by the ethical principles regarding medical research conducted on human subjects, as set out in the Declaration of Helsinki of the World Medical Association. In turn, it will act in accordance with the provisions of Law 14/2007, of July 3, on Biomedical Research.

Also, each participant will be given an informed consent form, prepared following Law 41/2002, which they must sign and in which, their voluntary participation in said study will be verified. Entry to the study is voluntary and the decision to participate or not will not affect the medical care or treatment of patients. Patients who are interested in participating in this study will be explained what it is and will be given the information sheet. Those who choose to join will sign the informed consent at the beginning of the study, approving the desire to take part on an ongoing basis and agreeing to be contacted throughout the study and follow-up process. They will also be informed about the possibility of leaving the study at any time without having to communicate the reason and without affecting their subsequent treatment/clinical follow-up.

Finally, the study will be carried out following the regulations of Law 15/99, of December 13, which aims to guarantee and protect, with regard to the processing of personal data, public freedoms and the fundamental rights of natural persons, and especially their honor and personal and family privacy.

ELIGIBILITY:
Inclusion Criteria:

* People from 18 to 65 years old
* Shoulder pain of at least three months of evolution located in the proximal anterolateral region of the shoulder
* Presenting shoulder pain during movements with a history of traumatic or insidious onset
* Agree to participate in the study and sign the informed consent

Exclusion Criteria:

* Shoulder pain resulting from a dysfunction of the cervical spine.
* Cognitive deficits
* Uso of medicines for pain control in the previous 24 hours,
* A history of neurological or psychiatric disorders
* Adhesive capsulitis syndrome (limited passive range of motion of the shoulder: external rotation < 30°; elevation < 150°)
* Patients with shoulder instability
* Previous surgery of the shoulder
* Rheumatic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-04 (Estimated); Primary Completion 2024-07-03 (Estimated); Study Completion 2024-07-03 (Estimated)

PRIMARY OUTCOMES:
Range of movement in flexion of the shoulder | Change from Baseline after the intervention up to 1 day
  Digital Goniometry: Scores 0-180 grades
Pain during shoulder flexion movement | Change from Baseline after the intervention up to 1 day
  Visual Analogue Pain Scale: scores 0-10

SECONDARY OUTCOMES:
Hand grip strength | Change from Baseline after the intervention up to 1 day
  Digital dynamometry: scores 0-1000 newtons
Pain Self-efficacy | Change from Baseline after the intervention up to 1 day
  Self-efficacy questionnaire in chronic pain: Score from 0 to 190
Disability | Change from Baseline after the intervention up to 1 day
  Questionnaire shoulder and pain disability index (SPADI-sp): Score from 0 to 130
Kinesiophobia | Change from Baseline after the intervention up to 1 day
  Tampa Questionnaire for Kinesiophobia (TSK-11): Score from 11 to 44
Age | Baseline
  Self-developed questionnaire
Sex | Baseline
  Self-developed questionnaire
Profession | Baseline
  Self-developed questionnaire
Marital Status | Baseline
  Self-developed questionnaire
Fear of pain | Change from Baseline after the intervention up to 1 day
  Pain fear questionnaire (FPQ-III): Score 0-150
Risk Chronicity | Change from Baseline after the intervention up to 1 day
  Örebro Musculoskeletal Pain Questionnaire (OMPQ): Score from 0-210

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad Docente Asistencial Fisioterapia, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Page MJ, O'Connor DA, Malek M, Haas R, Beaton D, Huang H, Ramiro S, Richards P, Voshaar MJH, Shea B, Verhagen AP, Whittle SL, van der Windt DA, Gagnier JJ, Buchbinder R; OMERACT Shoulder Core Set Working Group. Patients' experience of shoulder disorders: a systematic review of qualitative studies for the OMERACT Shoulder Core Domain Set. Rheumatology (Oxford). 2019 Mar 6:kez046. doi: 10.1093/rheumatology/kez046. Online ahead of print. PMID 30843587
- [Background] Meehan K, Wassinger C, Roy JS, Sole G. Seven Key Themes in Physical Therapy Advice for Patients Living With Subacromial Shoulder Pain: A Scoping Review. J Orthop Sports Phys Ther. 2020 Jun;50(6):285-a12. doi: 10.2519/jospt.2020.9152. PMID 32476583
- [Background] Farzad M, MacDermid JC, Ring DC, Shafiee E. A Scoping Review of the Evidence regarding Assessment and Management of Psychological Features of Shoulder Pain. Rehabil Res Pract. 2021 Sep 30;2021:7211201. doi: 10.1155/2021/7211201. eCollection 2021. PMID 34631168
- [Background] Martinez-Calderon J, Meeus M, Struyf F, Miguel Morales-Asencio J, Gijon-Nogueron G, Luque-Suarez A. The role of psychological factors in the perpetuation of pain intensity and disability in people with chronic shoulder pain: a systematic review. BMJ Open. 2018 Apr 13;8(4):e020703. doi: 10.1136/bmjopen-2017-020703. PMID 29654040
- [Background] Alaiti RK, Caneiro JP, Gasparin JT, Chaves TC, Malavolta EA, Gracitelli MEC, Meulders A, da Costa MF. Shoulder pain across more movements is not related to more rotator cuff tendon findings in people with chronic shoulder pain diagnosed with subacromial pain syndrome. Pain Rep. 2021 Dec 16;6(4):e980. doi: 10.1097/PR9.0000000000000980. eCollection 2021 Nov-Dec. PMID 34938935
- [Background] Mallari B, Spaeth EK, Goh H, Boyd BS. Virtual reality as an analgesic for acute and chronic pain in adults: a systematic review and meta-analysis. J Pain Res. 2019 Jul 3;12:2053-2085. doi: 10.2147/JPR.S200498. eCollection 2019. PMID 31308733
- [Background] Matamala-Gomez M, Donegan T, Bottiroli S, Sandrini G, Sanchez-Vives MV, Tassorelli C. Immersive Virtual Reality and Virtual Embodiment for Pain Relief. Front Hum Neurosci. 2019 Aug 21;13:279. doi: 10.3389/fnhum.2019.00279. eCollection 2019. PMID 31551731
- [Background] Lin I, Wiles L, Waller R, Goucke R, Nagree Y, Gibberd M, Straker L, Maher CG, O'Sullivan PPB. What does best practice care for musculoskeletal pain look like? Eleven consistent recommendations from high-quality clinical practice guidelines: systematic review. Br J Sports Med. 2020 Jan;54(2):79-86. doi: 10.1136/bjsports-2018-099878. Epub 2019 Mar 2. PMID 30826805